CLINICAL TRIAL: NCT05528185
Title: Family Participation in Cardiac Intensive Care Unit Rounds: A Randomized Controlled Trial (The FAM-CICU Study)
Brief Title: Family Participation in CICU Rounds: RCT
Acronym: FAM-CICU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lady Davis Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2022-3175
Record Dates: First submitted 2022-08-24; First posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-08

CONDITIONS: Family Members; Health Care Providers; Engagement, Patient
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Health care providers will be blinded to participants who are randomized to usual care.
  The investigator and outcomes assessor will be blinded to treatment assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention consists of family participation in morning interdisciplinary team rounds in the cardiac ICU. Family participation will consist of orientation, engagement, summary, questions, and communication follow-up by the care team.
  Interventions: Other: Direct participation of the family member in the daily rounds
- Usual care (No Intervention): Usual care consists of interdisciplinary team rounds that occur outside the patient's room each morning without a family member present.

INTERVENTIONS:
Other: Direct participation of the family member in the daily rounds — When the team arrives at the participating family member's room, the family member will be invited by a member of the healthcare team to come out of the room. The rounding team and structure will be the same as the usual care group with the following exceptions: (1) the family member will be invited to participate in the rounds outside their relative's room; (2) the family member will be provided with an orientation to the medical team members; (3) the family member will be allowed to engage and participate throughout the rounds; (4) at the end of the rounds, the team will summarize the patient's daily care plan; (5) the family member will be prompted to ask questions.
  Arms: Intervention

SUMMARY:
This is a single-center, unblinded, pragmatic randomized controlled trial comparing family participation in cardiac ICU team rounds with usual care. We will recruit 112 family members. The primary outcome will be family member care satisfaction. Secondary outcomes will include family mental health and care engagement. The beliefs, attitudes, and knowledge of healthcare providers, including medical trainees, about family participation in rounds will be evaluated prior to and following the intervention.

DETAILED DESCRIPTION:
This is a single-center (Jewish General Hospital), unblinded, pragmatic randomized controlled trial comparing family participation in the Cardiac Intensive Care Unit (CICU) team rounds with usual care.

Research team will recruit family members and health care providers in the Cardiac Intensive Care Unit (CICU) at the Jewish General Hospital. Family members will be randomized in a 1:1 ratio to either the intervention or usual care using the REDCap randomization module. The intervention consists of family invitation and participation in team rounds during the patient's stay in the CICU. Family may participate in-person or virtually. Usual care consists of interdisciplinary team rounds that occur outside the patient's room each morning without family presence.

A research team member will approach the participating family member to distribute the follow-up survey after transfer of the patient to the cardiovascular ward or prior to hospital discharge if the patient will be discharged from the hospital directly from the CICU. The follow-up survey will be composed of the FS-ICU, HADS, and FAME surveys. The perspectives of healthcare providers, including medical trainees, prior to and after the intervention will be assessed through the QFIFE survey.

An increase in the mean family care satisfaction score, as measured by the Family Satisfaction in the ICU survey (FS-ICU) is hypothesized for family members participating in team rounds. A positive change in attitudes and knowledge of healthcare providers and medical trainees following family participation in rounding is also expected.

The proposed study will generate much needed evidence for the effectiveness of a family rounding strategy to improve family-centered outcomes in the cardiac ICU. The evidence derived from this study could support the practice of family participation in team rounding and inform clinicians about the potential benefits of this approach.

ELIGIBILITY:
Inclusion Criteria:

* expected patient length of stay >48 hours
* family member, as designated by the patient or surrogate decision maker
* able to participate in English or French
* willingness to participate in morning rounds

Exclusion Criteria:

* another family member has already participated in the study
* inability to provide informed consent in English or French

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Family Care Satisfaction as Measured by the FS-ICU Survey. | Within 2 weeks of cardiac ICU discharge
  A mean improvement change in Family Satisfaction in the ICU (FS-ICU 24R) survey score in family members participating in rounds (intervention). The survey assesses family satisfaction with care in the ICU setting and is given at the end of the patient's stay in the Cardiac Intensive Care Unit. Survey scores are reported with a range of 0-100, where higher scores indicate increased satisfaction with care.

SECONDARY OUTCOMES:
Family Engagement in Care as Measured by the FAMily Engagement (FAME) Survey | Within 2 weeks of cardiac ICU discharge
  The survey assesses perception of engagement, family presence, communication/education, decision-making, contributing to care, family-centered care, and family needs. A five-point Likert scale is used for response. Scale results are then transformed to a 0-100 scoring system, with higher scores indicating greater engagement in care and lower scores indicating lesser engagement in care.
Family Mental Health as Measured by the Hospital Anxiety and Depression Scale (HADS) Survey | Within 2 weeks of cardiac ICU discharge
  The Hospital Anxiety and Depression Scale (HADS) is a self-reported tool to measure anxiety and depression in medical patients. It is composed of 14 questions (7 depression-related and 7 anxiety-related) on a 4-point Likert scale (range 0-3). The total score is the sum of the 14 questions, and for each subscale the score is the sum of the respective 7 questions.
Change in Attitudes and Knowledge of Healthcare Providers as measured by the QFIFE survey | Through study completion, up to 4 weeks
  The Questionnaire on Factors That Influence Family Engagement (QFIFE) assesses the perspectives of healthcare providers and medical trainees. Health care providers will take the QFIFE questionnaire (pre-intervention) prior to their first exposure to the intervention. At the end of the intervention period, participating health care providers will take the QFIFE questionnaire a second time (post-intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Goldfarb, MD,MSc, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Abdallah JP, Morel SBA, Soboleva N, Quan J, Price C, Goldfarb M. A Digital Tool to Improve Family Engagement in Acute Care: The NGAGE Randomized Pilot Feasibility Trial. CJC Open. 2025 Mar 11;7(6):743-749. doi: 10.1016/j.cjco.2025.03.007. eCollection 2025 Jun. PMID 40586017
- [Derived] Debay V, Hallot S, Calderone A, Goldfarb M. Family Participation in Cardiovascular Intensive Care Unit Rounds: A Pilot Randomized Controlled Trial. CJC Open. 2023 May 16;5(8):619-625. doi: 10.1016/j.cjco.2023.05.002. eCollection 2023 Aug. PMID 37720185